CLINICAL TRIAL: NCT01650610
Title: Gait Training Associated With Executive Functions Tasks in Subjects With Parkinson´s Disease: A Study Protocol
Brief Title: Gait Training With Executive Functions Tasks in Subjects With Parkinson´s Disease: A Study Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Cynthia Bedeschi Ferrari, PhD Student, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USPNEC001
Record Dates: First submitted 2012-07-19; First posted 2012-07-26 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson´s Disease
Keywords: Parkinson´s Disease; Rehabilitation; Cognition
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gait training executive functions tasks (Experimental): This group will perform a gait training associated with the tasks that require the main executive functions.
  Interventions: Behavioral: Gait training executive functions tasks

INTERVENTIONS:
Behavioral: Gait training executive functions tasks — The training will consist of 10 sessions, two times per week for five weeks, and consists of 30 minutes of global exercises that involves stretching, muscle strengthen and axial mobility exercises, and another 30 minutes of gait training in a dual-task condition associated with distracting tasks that require handling of the main executive functions: volition, self-awareness, planning, response inhibition, response monitoring and attention.

SUMMARY:
The aim of this study is the development and implementation of a new protocol of a physical therapy training, based on a gait training associated with executive tasks, for treatment of individuals with Parkinson's Disease.

The hypothesis is that this group of patients who will carry out training of this study protocol will show improvement in measured parameters (functionality of gait and cognitive ability), which allows this protocol to be improved and published as a proposal of physiotherapeutic treatment.

DETAILED DESCRIPTION:
The aim of this study is the development and implementation of a new protocol of physical therapy training, based on a gait training associated with executive tasks for treatment of individuals with Parkinson's Disease.

The proposed motor training consists of 30 minutes of global exercises that involves stretching, muscle strengthen and axial mobility exercises, and after this, 30 minutes of gait training in a dual-task condition, associated with distracting tasks that require handling of the main executive functions.

It will be an open label study, non randomized, where 30 patients with PD in stages 1 to 3 on Hoehn & Yahr scale will participate in the study, to be held in Brazil Parkinson Association. The training will consist of 10 sessions, two times per week for five weeks.

The executive tasks concomitant with gait training cover the following executive functions: volition, self-awareness, planning, response inhibition, response monitoring and attention.

The main outcome measures are: (1) Dynamic Gait Index (DGI), (2) Montreal Cognitive Assessment (MoCA), (3) Trail Making Test A and B, (4) Unified Parkinson's Disease Rating Scale (UPDRS) and (5) Falls Efficacy Scale (FES).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic PD performed by a neurologist specialist in movement disorders;
* In use of dopaminergic medication;
* Disease severity of 1 to 3 according to Hoehn & Yahr scale;
* Absence of other neurological disorders or co-morbidities that may affect gait;
* Absence of dementia (score above 24 on the Mini Mental State Examination - MMSE);
* Vision and hearing adequate or corrected to normal;
* Ability to walk independently;
* Absence of prolonged off state;
* Age 50 to 85 years.

Exclusion Criteria:

* Biomechanical alterations (other pathologies) that could compromise the completion of training;
* Presence of depression, detected by the Geriatric Depression Scale (GDS-15);
* Presence of any neurological, auditory or visual deficit that could compromise distracting task performance during gait training;
* Any changes in drug treatment for PD.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-02 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Index | 02/2013 (Up to seven months)
  The scale assesses the ability to adapt the gait during motor tasks with different demands.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | 02/2013 (Up to seven months)
  This scale was developed in order to detect mild degrees of cognitive impairment. The instrument assesses different cognitive domains such as attention and concentration, executive functions, memory, language, visuo-constructive skills, calculations, and orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PhD, Study Director — University of Sao Paulo; Cynthia B Ferrari, PhD Student, Principal Investigator — University of Sao Paulo
Locations (1):
- Brazil Parkinson Association, São Paulo, São Paulo, Brazil